CLINICAL TRIAL: NCT00880594
Title: The Modulation of Cerebral Pain Responses Using Desipramine in the Treatment of Irritable Bowel Syndrome (IBS)
Brief Title: Irritable Bowel Syndrome (IBS) Functional Magnetic Resonance Imaging (fMRI) With Desipramine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to changes in trial personnel (co-investigator and research coordinator leaving the institution).
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-0013
Record Dates: First submitted 2009-04-13; First posted 2009-04-14 (Estimated); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Desipramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IBS-High somatization (Experimental): Participants meeting Rome III criteria for IBS and with high somatization (PHQ≥10)
  Interventions: Drug: Desipramine
- IBS-Low somatization (Experimental): Participants meeting Rome III criteria for IBS and with high somatization (PHQ≤5)
  Interventions: Drug: Desipramine

INTERVENTIONS:
Drug: Desipramine — Desipramine 25 mg/day administered in the evening. Dosing may be increased dependent upon side-effects and clinical response to a maximum of 100 mg/day. Absent significant side-effects, all patients are increased at the one week visit to 50 mg/day at bedtime if they have not achieved a report of "Adequate relief". Thereafter, up to week 4, the daily desipramine dose may be increased weekly by 25 mg up to the 100 mg/d maximum.

SUMMARY:
Individuals with irritable bowel syndrome (IBS) may experience abdominal pain as a result of pain signals in the bowel and how these signals are processed in the brain. Studies using brain imaging (pictures) have shown that IBS patients with more pain diagnoses (i.e. fibromyalgia, migraines, etc.) have greater activity in the regions of the brain responsible for the emotional and thought processing of pain signals. This could possibly make bowel sensations and bowel difficulties feel abnormal or more noticeable, in turn causing more severe IBS symptoms. The purpose of this protocol is to explore the role of pain diagnoses and their affect on brain activity in IBS patients. The investigators will also examine the use of a medication, desipramine, which is known to affect these brain regions, in IBS patients.

DETAILED DESCRIPTION:
Background Irritable bowel syndrome (IBS) is a common abdominal pain disorder diagnosed by symptom-based criteria (Rome III). Since there is no objective measure available to establish a formal diagnosis, IBS likely encompasses a biologically heterogeneous group of patients with distinct pathophysiology. To date, studies evaluating the mechanistic basis of IBS largely have focused on bowel-specific factors. More recently, differences in brain activation patterns in response to painful visceral stimuli (rectal balloon distention) have been identified in IBS subjects compared to healthy controls. These differences often are observed within the homeostatic afferent processing network (HAPN), regions of the brain responsible for the descending inhibition of pain signals, as well as the affective and emotional response to pain. However, IBS brain activation patterns are inconsistent across IBS studies. One likely explanation for this variation in brain activations is the role of psychiatric co-morbidity often present in IBS. No study to-date has considered whether unique patterns of cerebral activation during visceral stimulation exist among subgroups of IBS patients. In our current work, we are exploring the role of multiple co-morbid unexplained pain syndromes, hereafter referred to as 'somatization', and its relevance to IBS subjects' brain responses to pain. We anticipate that IBS patients with somatization (IBS-S+) have aberrant descending inhibitory neurocircuitry, facilitating more intense pain experiences across a spectrum of ascending pain signals (both visceral and somatic). Somatization can be readily detected using standardized instruments and medical histories, and when present in IBS subjects clinically portends more severe bowel symptoms, and poorer responses to proven bowel-specific IBS therapies. Greater insight into the relevance of somatization and mood symptoms to HAPN brain networks thus is not only critical to our understanding of the pathophysiology of IBS, but also may reveal additional clinical targets for the management of these disorders.

Hypotheses and Aims The overarching hypothesis of this proposal is that abnormal homeostatic afferent processing network (HAPN) responses to visceral stimulation have mechanistic relevance to a subset of patients with IBS. It is further hypothesized that abnormalities HAPN responses to afferent pain signals in IBS subjects with comorbid somatization (IBS-S+) result in: (1) more generalized pain experiences (both visceral and somatic), and (2) more severe IBS and somatic pain symptom experiences.

Using functional magnetic resonance imaging (fMRI), our preliminary findings have revealed abnormal activation of HAPN brain regions following visceral stimulation in IBS subjects compared to healthy controls. Our pilot data also demonstrated a distinct pattern of abnormal HAPN activations in response to visceral stimulation in IBS subjects with comorbid somatization (IBS-S+) compared to those without somatization (IBS-S-). These findings suggest that clinical differences between IBS-S+ and IBS-S- subjects may result from aberrant HAPN responses to visceral sensory input. The purpose of this proposal is to further investigate the mechanistic importance of the brain's homeostatic afferent processing network in the presence of overlapping somatization and mood disorders to symptom experiences in IBS.

This goal will be realized through the pursuit of the following Specific Aims:

Specific Aim 1. To validate homeostatic afferent processing network (HAPN) activation patterns with noxious visceral stimulation in IBS subjects, and determine their relationship to visceral pain symptom experiences.

Hypothesis 1: IBS subjects collectively will demonstrate a pattern of abnormal HAPN activation in response to noxious visceral stimulation Hypothesis 1b: Abnormal HAPN brain activations overall will correlate with greater subjective pain ratings of noxious visceral stimulation in IBS subjects Specific Aim 2. To evaluate the influence of somatization on HAPN activations with noxious visceral and somatic stimulation in IBS subjects, and determine their relationship to pain symptom experiences.

Hypothesis 2: IBS subjects with comorbid somatization (IBS-S+) will demonstrate abnormal HAPN activation in response to both noxious visceral and somatic stimuli, when compared to IBS subjects with no somatization (IBS-S-).

Specific Aim 3: To determine the influence of despiramine on abnormal HAPN brain activations in IBS-S+ and IBS-S- subjects.

Hypothesis 3: Desipramine will normalize HAPN activations in both IBS-S+ and IBS-S-, with greater effects in the IBS-S+ cohort.

ELIGIBILITY:
Inclusion Criteria:

* IBS subjects with- and without comorbid somatization features will be recruited from the sources highlighted above.
* To be eligible, subjects will have to be between 18 and 90 years of age (inclusive) and qualify for a diagnosis of irritable bowel syndrome according to the criteria set forth in the Rome III criteria for the Diagnosis of Functional GI Disorders.
* IBS patients will then be assessed in terms of comorbid somatization as determined using the Patient Health Questionnaire-15 (PHQ-15).
* For this particular study, only subjects with high somatization (PHQ ≥ 10 or low somatization (PHQ ≤5) will be considered for enrollment.
* Verification of somatization status will be performed using a formal structured interview process (Diagnostic Interview Schedule, DIS).
* Persons are eligible to participate without regard to race or ethnicity.
* Given sex differences in cerebral responses to noxious stimuli and the greater prevalence of IBS in women, only female participants will be sought in this study.
* Also, in view brain hemispheric differences between left- and right-hand dominant individuals and the greater prevalence of right-handedness, all participants must be right-handed

Exclusion Criteria:

* Persons are excluded from participation for having various psychiatric, medical, and other characteristics.
* Psychiatric/cognitive exclusions include any of the following: active suicidal or homicidal ideation or a history of attempted suicide, current excessive alcohol use or other substance abuse disorders, active major depression, anxiety disorder, bipolar depression or any psychotic disorder, unwillingness to be randomized or provide informed consent, inability to communicate with staff or significant cognitive impairment.
* Medical and other exclusions include any of the following: renal or hepatic disease or impairment, diabetes, cardiovascular disease, cardiac arrythmia, cerebrovascular disease, or breastfeeding, pregnant, or imminent intention of pregnancy, history of seizures or primary neurological disorder, head trauma, brain damage, hyper- or hypothyroidism, history or abdominal surgery (other than cholecystectomy/appendectomy), or known structural GI disorder (Crohn's disease, etc.), contraindication to MRI (metallic implant, pacemaker), or rectal balloon distention (e.g., proctitis/colitis).
* Exclusions related to medications:

  1. Analgesics (narcotics, NSAIDs; acetaminophen OK)
  2. Muscle relaxants
  3. Psychoactive agents (antidepressants, antipsychotics)
  4. Other medications (phenytoin; amphetamines, prescription weight-loss drugs, or benzodiazepines)
  5. Thyroid medication
  6. Anticholinergic medications or other IBS medications (hyoscyamine, dicyclomine)
  7. Cytochrome p450 substrates
  8. Participation in any clinical trial using any other drug.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-02; Primary Completion 2014-11-11 (Actual); Study Completion 2014-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory S. Sayuk, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- IBS-High Somatization (Open Label Desipramine): IBS patients with high somatization (IBS-S+, ) IBS defined by Rome III, somatization by high PHQ-15.
  Desipramine: Desipramine 25 mg/day administered in the evening. Dosing may be increased dependent upon side-effects and clinical response to a maximum of 100 mg/day. Absent significant side-effects, all patients are increased at the one week visit to 50 mg/day at bedtime if they have not achieved a report of "Adequate relief". Thereafter, up to week 4, the daily desipramine dose may be increased weekly by 25 mg up to the 100 mg/d maximum.
- IBS-Low Somatization (Open Label Desipramine): IBS patients with low somatization (IBS-S-, ) IBS defined by Rome III, somatization by low PHQ-15 Desipramine: Desipramine 25 mg/day administered in the evening. Dosing may be increased dependent upon side-effects and clinical response to a maximum of 100 mg/day. Absent significant side-effects, all patients are increased at the one week visit to 50 mg/day at bedtime if they have not achieved a report of "Adequate relief". Thereafter, up to week 4, the daily desipramine dose may be increased weekly by 25 mg up to the 100 mg/d maximum.
Period: Overall Study
Arm/Group | IBS-High Somatization (Open Label Desipramine) | IBS-Low Somatization (Open Label Desipramine)
Started | 10 | 8
Completed | 5 | 4
Not Completed | 5 | 4
Not completed — Subject did not initiate desipramine therapy | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IBS-High Somatization | IBS-Low Somatization | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (13.65) | 42.38 (14.05) | 42.84 (13.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 9 | 5 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: MRI Blood Oxygen Level Dependent (BOLD) Activation CONTRASTS (in Prespecified Regions of Interest (ROI) in VOXELS
Description: CONTRASTS (comparisons of study group BOLD activations vs rest) are the outcome of interest. Voxel-wise comparisons (ANOVAs) were performed to determine differences in activations between groups within these regions. First level analyses of rectal balloon distensions experienced by subjects were modeled as box car functions then convolved with the canonical hemodynamic response function (HRF). For the second level analyses, differences in brain activation while experiencing both high and low painful rectal balloon distensions between IBS patients with High somatization vs Low somatization were examined with two-sample t-tests utilizing contrast images generated from the first level analysis. Unconventionally, these inferential statistics are regarded as the primary outcome in the study. Accordingly individual group level BOLD values where not recorded or evaluated separately in the cohorts. These data are not available, and cannot be reported "per Arm".
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: arbitrary unit
Groups:
- IBS-High Somatization: IBS patients with elevated PHQ-15
- IBS-Low Somatization: IBS patients with normal PHQ-15
Arm/Group | IBS-High Somatization | IBS-Low Somatization
Number analyzed (Participants) | 10 | 8
arbitrary unit
  Left insula activation contrast, Montreal Neurological Institute x,y,z coordinates (-28.5, 9, 19.5) | 0.02 (0.045) | -0.09 (0.07)
  Right insula activation contrast, Montreal Neurological Institute x,y,z coordinates (27, -1.5, 15) | 0.02 (0.04) | -0.09 (0.06)

ADVERSE EVENTS:
Time Frame: 1 month of treatment
Description: Per clinicaltrials.gov definitions
Groups:
- IBS-High Somatization: IBS patients with PHQ-15 ≥10
- IBS-Low Somatization: IBS patients with PHQ-15 ≤5
- Healthy Controls: Patients without IBS
Arm/Group | IBS-High Somatization | IBS-Low Somatization | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/15
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/15

LIMITATIONS AND CAVEATS:
Desipramine open-label completion target not achieved

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-08-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT00880594/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT00880594/ICF_001.pdf